CLINICAL TRIAL: NCT02762890
Title: Comparison of Deep Neuromuscular Block and Moderate Neuromuscular Block on Quality of Recovery in Patients Undergoing Robotic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2016-0206
Record Dates: First submitted 2016-05-04; First posted 2016-05-05 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep neuromuscular blockade (Experimental): Rocuronium will be administered continuously to achieve post-tetanic count 1-2 during surgery.
  Interventions: Drug: Deep neuromuscular blockade
- Moderate neuromuscular blockade (Active Comparator): Rocuronium will be administered continuously to achieve Train-of-four 1-2 during surgery.
  Interventions: Drug: Moderate neuromuscular blockade

INTERVENTIONS:
Drug: Deep neuromuscular blockade — neuromuscular blockade will be performed using a continuous infusion of rocuronium. Post-tetanic count 1-2 will be maintained during surgery. After the end of surgery, sugammadex of 4 mg/kg will be administered to reverse neuromuscular blockade.
  Arms: Deep neuromuscular blockade
Drug: Moderate neuromuscular blockade — neuromuscular blockade will be performed using a continuous infusion of rocuronium. Train-of-four 1-2 will be maintained during surgery. After the end of surgery, sugammadex of 2 mg/kg will be administered to reverse neuromuscular blockade.
  Arms: Moderate neuromuscular blockade

SUMMARY:
The purpose of this study is to investigate and compare the postoperative quality of recovery between the deep neuromuscular blockade and moderate neuromuscular blockade during robotic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 19-80 years who are scheduled for robotic gastrectomy

Exclusion Criteria:

* Neuromuscular disease
* History of malignant hyperthermia
* Significant renal or hepatic dysfunction
* Allergy to sugammadex or rocuronium

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Postoperative quality of recovery | within 48 hours after the end of surgery.
  The postoperative quality of recovery will be evaluated at 24 and 48 hours after the end of surgery by the investigator who are blinded to the group assignments.

SECONDARY OUTCOMES:
Surgical condition | within 48 hours after the end of surgery
  Surgical condition will be evaluated after the end of surgery by the investigator who are blinded to the group assignments.
shoulder pain | within 48 hours after the end of surgery
  shoulder pain will be evaluated after the end of surgery by the investigator who are blinded to the group assignments.
abdominal pain | within 48 hours after the end of surgery
  abdominal pain will be evaluated after the end of surgery by the investigator who are blinded to the group assignments.
nausea and vomiting | within 48 hours after the end of surgery
  nausea and vomiting will be evaluated after the end of surgery by the investigator who are blinded to the group assignments.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data